CLINICAL TRIAL: NCT04620278
Title: Genetic Investigation of Cancer Predisposition
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: HSC20200666H
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Genetic Predisposition; Cancer
Keywords: Genetic analysis; Early diagnosis
MeSH Terms: conditions — Genetic Predisposition to Disease; Neoplasms; Disease | interventions — DNA; Sequence Analysis, RNA

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: DNA or RNA Sequencing — Samples will be used for whole exome (DNA) or RNA sequencing

SUMMARY:
Clinical information and samples (blood, saliva, and tumor) will be collected from patients with multiple cancers and/or a family history of cancer as well as from affected and unaffected relatives; samples will be systematically sequenced and evaluated for candidate driver mutations.

DETAILED DESCRIPTION:
Genetic screening will be performed on DNA (and/or RNA) isolated from collected samples from affected individuals by whole exome sequencing or RNA sequencing using in-house pipeline to identify candidate sequence variants. These variants will be tested for segregation with the phenotype in other relatives (affected/unaffected). Candidate variants will be subjected to additional downstream analysis, to be guided by the actual type of gene/variant.

ELIGIBILITY:
Inclusion Criteria:

1. Any age
2. Meets at least ONE of the following:

   1. Personal history (with documented diagnosis) of cancer before the age of 50
   2. Personal history of more than one primary cancer
   3. Documented diagnosis of cancer AND family history of that same cancer type or multiple other cancers that do not fit classical criteria of hereditary cancer syndromes
   4. Documented diagnosis of a rare cancer AND family history of rare cancers that do not fit classical criteria of hereditary cancer syndromes
   5. There is the same type of cancer in several generations of a family
   6. Documented diagnosis of multicentric cancers (e.g bilateral cancers in paired organs, or multifocal cancers in single organs) that usually occur as single lesions when presented sporadically
   7. Early onset cancer (before the age of 50, or breast cancer before age 45) AND family history of early onset cancer Capable of providing access to detailed medical records and family history of cancer

Exclusion Criteria:

1. Established genetic diagnosis of a known hereditary cancer syndrome that is compatible with the clinical presentation
2. Incarcerated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a family history of cancer or with a personal history of multiple cancers that might suggest increased genetic predisposition, but for which an identifiable susceptibility mutation has not been detected.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Identification of Rare Genetic Variant | through study completion- approximately 6-12 months
  Genetic screen detects a mutation that is likely responsible for tumor development
Identification of somatic (tumor only) mutation | through study completion- approximately 6-12 months
  Genetic screen detects a mutation that is likely responsible for tumor development
Identification of Rare Genetic Variant in family members | through study completion- approximately 6-12 months
  Genetic screen detects a mutation that is likely responsible for tumor development

SECONDARY OUTCOMES:
Identification of clinical spectrum of the disease in families | through study completion- approximately 6-12 months
  Genetic and clinical analysis reveals clinical features not previously assigned to the disease

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Dahia, MD, PhD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All information exchanged between the local investigator/referring physician and the PI will be made through the unique identifiers to maintain patient confidentiality
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the age-related penetrance of the disease is not known, it may be many years before an individual changes his/her affection status. Thus, the clinical updates remain open-ended
Access Criteria: PI will provide coded data to collaborators who have signed an MTA agreement. These collaborators will not have access to identifiable data